CLINICAL TRIAL: NCT00592384
Title: A Controlled Trial of Venlafaxine XR for Major Depression After Spinal Cord Injury: A Multi-site Study
Brief Title: Project to Improve Symptoms and Mood in People With Spinal Cord Injury
Acronym: PRISMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Michigan (Other); Shirley Ryan AbilityLab (Other); University of Alabama at Birmingham (Other); Baylor Health Care System (Other); University of Miami (Other); New York University (Other)
Responsible Party: Principal Investigator, Charles Bombardier, Primary Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31665-D; H133A060107; (Other Grant/Funding Number: National Institute on Disability and Rehabilitation Research)
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Major Depressive Disorder; Dysthymia; Spinal Cord Injuries
Keywords: spinal cord injuries; major depressive disorder; dysthymia; antidepressant agents; pain; quality of life; muscle spasticity; community participation; anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Spinal Cord Injuries; Pain; Muscle Spasticity; Anxiety Disorders | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): identically encapsulated placebo pills 37.5 - 300 mg/day for 12 weeks
  Interventions: Drug: placebo
- venlafaxine XR (Experimental): venlafaxine XR 37.5 - 300 mg/day for 12 weeks
  Interventions: Drug: venlafaxine XR

INTERVENTIONS:
Drug: venlafaxine XR — Once daily oral dose of venlafaxine XR ranging from 37.5 mg up to 300 mg
  Other Names: Effexor XR
  Arms: venlafaxine XR
Drug: placebo — Once daily oral dose of placebo ranging from 37.5 mg up to 300 mg
  Other Names: identically encapsulated inactive substance
  Arms: placebo

SUMMARY:
Depression is likely the most prevalent and disabling psychological complication associated with spinal cord injury (SCI). Yet no controlled depression treatment trials have been performed in this population. The proposed study is a multi-site, randomized, double-blind, placebo controlled trial of venlafaxine XR (Effexor XR) in 133 adults with SCI and major depressive disorder (MDD) or dysthymia who are at least one month post injury. Participants will be recruited from four SCI Model System sites, the University of Washington, Rehabilitation Institute of Chicago, University of Michigan, University of Alabama, Birmingham and Baylor Institute for Rehabilitation, Dallas, TX. The purpose of the study is to examine the efficacy and tolerability of venlafaxine XR as a treatment for MDD. The primary outcome will be the percent of responders (those who report at least a 50% reduction in depression severity from baseline to the end of treatment) in the venlafaxine XR versus placebo control group using intent-to-treat analysis. Secondary outcomes will include changes in pain, health related quality of life depression-related disability and community participation. A successful clinical trial could lead to more aggressive identification and treatment of MDD as well as improved health and quality of life in this important population.

DETAILED DESCRIPTION:
Depression is likely the most prevalent and disabling psychological complication associated with spinal cord injury (SCI). The prevalence of major depression in people with SCI is 22% or two to six times higher than in the general population. Depression is linked to a myriad of adverse outcomes including poor subjective health, poor community integration, higher rates of medical complications and high rates of suicide. Surprisingly there are no randomized controlled trials for treating major depressive disorder (MMD) in people with SCI. Despite the widespread use of antidepressants in this population, the common assumption that antidepressant medications are effective and well-tolerated among people with SCI is uncertain. Multiple factors such as severe stresses, bereavement and loss of rewarding activities may complicate treatment. Treatment trials suggest antidepressants may not be as effective in people with medical/neurological conditions as they are with depression that develops as a primary condition. For almost 20 years clinicians and scientists have called for controlled clinical trials of antidepressants among people with SCI in order to establish evidence-based treatment. The proposed study is a multi-site, randomized, double-blind, placebo controlled trial of venlafaxine XR (Effexor XR) in 133 adults with SCI and MDD or dysthymia who are at least one month post injury. Participants aged 18-64 will be recruited from four SCI Model System sites, the University of Washington, Rehabilitation Institute of Chicago, University of Michigan, University of Alabama, Birmingham and Baylor Institute for Rehabilitation, Dallas TX. The purpose of the study is to examine the efficacy and tolerability of venlafaxine XR as a treatment for MDD. The primary outcome will be the percent of responders (those who report at least a 50% reduction in depression severity from baseline to the end of treatment) in the venlafaxine XR versus placebo control group using intent-to-treat analysis. Secondary outcomes will include changes in pain, health related quality of life and participation. A successful clinical trial could lead to more aggressive identification and treatment of MDD as well as improved health and quality of life in this important population.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (ASIA A-D)
* At least one month post injury
* Meets DSM IV criteria for major depression or dysthymia on the SCID
* At least moderately severe depression (PHQ-9 score >= 10)
* Within reasonable travel distance to one of the study sites

Exclusion Criteria:

* Current DSM IV alcohol or drug dependence
* History of bipolar disorder or psychosis
* History of >= 2 suicide attempts or suicide attempt with 5 years
* Current suicidal intent or plan
* Medical contraindications
* Non-English speaker
* Clinically significant cognitive/language impairment
* History of allergic reaction to venlafaxine XR or use of MAO-I with 2 weeks
* Current use of antidepressant medications (will not exclude if on low dose of a tricyclic antidepressant or trazodone for pain, sleep, or bladder), psychotherapy for depression, or electroconvulsive therapy
* Pregnant or lactating women or women of childbearing potential who are not willing to use a reliable form of contraception
* Unstable medical condition, as determined by physical examination, CBC w/ platelets (including hematocrit, hemoglobin, WBC, differential), serum chemistry panel (serum sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose), liver transaminases (AST, ALT), thyroid stimulating hormone (TSH), urinalysis, supine diastolic blood pressure (SDBP) > 90 mm Hg, or near terminal illness (primary care physician estimates that patient has < 1 year to live)
* Anticipated major surgical procedures within the 12 weeks of randomization
* Use of an investigational drug within 30 days
* Use of psychoactive medications, including corticosteroids and anticonvulsants, that have not been at a stable dose for at least 2 weeks
* Use of anxiolytic, sedative-hypnotic, or other psychotropic drug or substance (including St. John's Wort) within 7 days of start of double-blind treatment. If the patient is taking a sedative deemed necessary for sleep induction or spasticity, the dosage must have been stable for at least 2 weeks. Use of anticholinergic, low-dose tricyclic antidepressant, GABAergic or adrenergic medications for spasticity are permitted if at a stable dose for at least 2 weeks.
* Refusal to participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H. Bombardier, PhD, Principal Investigator — University of Washington School of Medicine, Department of Rehabilitation Medicine; Jesse R. Fann, MD, MPH, Principal Investigator — University of Washington School of Medicine, Department of Psychiatry and Behavioral Science
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Baylor Institute for Rehabilitation, Dallas, Texas
  - University of Washington/Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] McCullumsmith CB, Kalpakjian CZ, Richards JS, Forchheimer M, Heinemann AW, Richardson EJ, Wilson CS, Barber J, Temkin N, Bombardier CH, Fann JR; PRISMS Investigators. Novel risk factors associated with current suicidal ideation and lifetime suicide attempts in individuals with spinal cord injury. Arch Phys Med Rehabil. 2015 May;96(5):799-808. doi: 10.1016/j.apmr.2014.12.017. Epub 2015 Jan 19. PMID 25613597
- [Derived] Fann JR, Bombardier CH, Richards JS, Wilson CS, Heinemann AW, Warren AM, Brooks L, McCullumsmith CB, Temkin NR, Warms C, Tate DG; PRISMS Investigators. Venlafaxine extended-release for depression following spinal cord injury: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):247-58. doi: 10.1001/jamapsychiatry.2014.2482. PMID 25607727
- [Derived] Bombardier CH, Fann JR, Tate DG, Richards JS, Wilson CS, Warren AM, Temkin NR, Heinemann AW; PRISMS Investigators. An exploration of modifiable risk factors for depression after spinal cord injury: which factors should we target? Arch Phys Med Rehabil. 2012 May;93(5):775-81. doi: 10.1016/j.apmr.2011.12.020. Epub 2012 Mar 20. PMID 22440484
- [Derived] Fann JR, Bombardier CH, Richards JS, Tate DG, Wilson CS, Temkin N; PRISMS Investigators. Depression after spinal cord injury: comorbidities, mental health service use, and adequacy of treatment. Arch Phys Med Rehabil. 2011 Mar;92(3):352-60. doi: 10.1016/j.apmr.2010.05.016. Epub 2011 Jan 20. PMID 21255766

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control: placebo: identically encapsulated inactive substance
- Venlafaxine XR: venlafaxine XR: Once daily oral dose ranging from 37.5 mg up to 300 mg
Period: Overall Study
Arm/Group | Placebo Control | Venlafaxine XR
Started | 64 | 69
Completed | 59 | 63
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control | Venlafaxine XR | Total
Number analyzed (Participants) | 64 | 69 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12) | 39 (11) | 40 (12)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 69 | 133
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 34
  Male | 51 | 48 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 19 | 42
  White | 38 | 48 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 55 | 64 | 119
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale-17
Description: The 17-item Hamilton Depression Rating Scale is a clinician rated measure of depression severity (we used a structured interview version (Williams 1988) to improve inter-rater reliability). Scores range from 0-52. Higher scores indicate more severe depression. Scores of 7 or less indicate remission from depression.
Time Frame: 0 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Control | Venlafaxine XR
Number analyzed (Participants) | 64 | 69
units on a scale
  Baseline | 19.5 (5.4) | 19.4 (5.5)
  12-week outcome | 9.5 (6.5) | 9.5 (7.3)
Statistical Analysis 1: Comparison: Placebo Control vs Venlafaxine XR; Primary analyses included observations at baseline, 1, 3, 6, 8, 10, and 12 weeks. Random effects were included for participants' intercepts. Fixed effects were time (linear), treatment (VFN vs. PBO), interaction of time with treatment, stratification factors and potential confounders and variables to improve sensitivity. The primary indicator of treatment effect was the interaction of time by treatment; Test type: Superiority or Other; p < .025, Mixed Models Analysis — Bonferroni corrected for two primary comparisons; see above

2. Secondary Outcome: Symptom Checklist-20 Depression Subscale
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12, 24
Reporting Status: Not Posted

3. Secondary Outcome: Modified Brief Pain Inventory
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12
Reporting Status: Not Posted

4. Secondary Outcome: Modified Ashworth Spasticity Scale
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12
Reporting Status: Not Posted

5. Secondary Outcome: Structured Clinical Interview for DSM IV Depression Module
Time Frame: Weeks 0, 12, 24
Reporting Status: Not Posted

6. Secondary Outcome: SF-12
Time Frame: Weeks 0, 12, 24
Reporting Status: Not Posted

7. Secondary Outcome: Side Effects Checklist
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12
Reporting Status: Not Posted

8. Secondary Outcome: Craig Handicap and Reporting Technique
Time Frame: Weeks 0, 12
Reporting Status: Not Posted

9. Secondary Outcome: Satisfaction With Life
Time Frame: Weeks 0, 12
Reporting Status: Not Posted

10. Secondary Outcome: Sheehan Disability Scale
Time Frame: Weeks 0, 12
Reporting Status: Not Posted

11. Secondary Outcome: Clinical Global Impression
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12
Reporting Status: Not Posted

12. Secondary Outcome: Patient Global Impression
Time Frame: Weeks 0, 1, 3, 6, 8, 10, 12
Reporting Status: Not Posted

13. Secondary Outcome: Hamilton Rating Scale for Anxiety
Time Frame: Weeks 0, 12
Reporting Status: Not Posted

14. Primary Outcome: Hamilton Depression Rating Scale-Maier Subscale
Description: The Maier is a 6-item sub scale of the Hamilton derived from Rasch analysis. It is a unidimensional scale with superior sensitivity to change. It excludes somatic items and is therefore especially appropriate for individuals who have substantial physical impairment and medical comorbidity. Scores can range from 0-22 with higher scores indicating more severe depression. Scores of 4 or less indicated in remission from depression.
Time Frame: 0 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Control | Venlafaxine XR
Number analyzed (Participants) | 64 | 69
units on a scale
  Baseline | 8.7 (2.8) | 9.1 (2.9)
  12-week outcome | 3.9 (3.5) | 3.5 (3.6)
Statistical Analysis 1: Comparison: Placebo Control vs Venlafaxine XR; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .025, Mixed Models Analysis — Bonferroni corrected for two primary outcomes

ADVERSE EVENTS:
Time Frame: Data were collected at each interim visit (weeks 1, 3, 6, 8, 10) and at the final outcome point (12 weeks)
Arm/Group | Placebo Control | Venlafaxine XR
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/69
Other Adverse Events (participants affected / at risk) | 5/64 | 2/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control (N=64) | Venlafaxine XR (N=69)
self-harm (Injury, poisoning and procedural complications) | 0 | 1 — Subject had self-inflicted knife wound to abdomen
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control (N=64) | Venlafaxine XR (N=69)
urinary tract infection (Renal and urinary disorders) | 2 | 0
heart palpitations (Cardiac disorders) | 0 | 1
urinary tract infection and pressure ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
blurry vision (Eye disorders) | 1 | 0
increased risk of suicide (Psychiatric disorders) | 1 | 0
increased spasticity (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less